CLINICAL TRIAL: NCT04104087
Title: The Effect of the Tunneling Technique With Subepithelial Connective Tissue Graft Versus Tunneling Technique With Deepithelialized Free Gingival Graft on the Papillary Height in the Treatment of RT2 Recession Defect: a Randomized Clinical Trial.
Brief Title: Comparing Deepithelialized Free Gingival Graft Versus Subpithelial Connective Tissue Graft With Tunneling Technique in Treating RT2 Gingival Recession
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Elshourbagy, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio 331
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: RT2 Gingival Recession
Keywords: tunneling technique, gingival recession, deepithelialized free gingival graft, sub epithelial connective tissue graft,
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: it is randomized control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deepithelializ free gingival graft (Experimental): performing tunneling technique with deepithelialized free gingival graft in treating RT2 gingival recession
  Interventions: Procedure: tunneling technique with sub epithelial connective tissue graft or deepithelialized free gingival graft.
- subepithelial connective tissue graft (Active Comparator): performing tunneling technique with sub epithelial connective tissue graft in treating RT2 gingival recession
  Interventions: Procedure: tunneling technique with sub epithelial connective tissue graft or deepithelialized free gingival graft.

INTERVENTIONS:
Procedure: tunneling technique with sub epithelial connective tissue graft or deepithelialized free gingival graft. — enhancing papillary hight and treating gingival recession RT2 by performing tunneling technique with sub epithelial connective tissue graft or deepithelialized free gingival graft.
  Other Names: root coverage

SUMMARY:
Complete coverage of the recession complemented with pleasing esthetics and minimal probing measures are the main goals of root coverage procedures.

According to a consensus report from the AAP regeneration workshop on the periodontal soft tissue root coverage procedures; most studies have been directed on RT-1 (Miller Class I and II) defects and that further research on results in RT-2, RT-3 ( Miller Class III and IV) defects is needed. Consequently, it was planned to conduct this research on RT-2 (Miller Class III) recessions to overcome this gap of knowledge, de-epithelialized free gingival graft is proposed aiming to enhance the papillary height, esthetic, with less pain and postoperative trauma. Equally, it is considered a more conservative approach with fewer complications.

DETAILED DESCRIPTION:
Gingival recession has high prevalence among both individuals with periodontal disease and those with high standers of oral hygiene. The management of RT-2 ( Miller Class III) gingival recessions is very challenging and there is controversy in the literature concerning the most predictable approach to treat these defects.

Treatment of gingival recession is performed to enhance esthetics, reduce dentinal hypersensitivity, eliminate caries risk, stop the progression of gingival recession and periodontal attachment loss and keratinized tissue augmentation to enable the patient to maintain adequate plaque control.Gingival recession or "Marginal tissue recession" is recognized as the apical migration of the marginal gingiva to its normal position on the root surface. Connective tissue graft (CTG) is considered to be the best root coverage techniques for the treatment of gingival recession defects.

However, it is challenging sometimes to harvest the largest volume of tissue especially in thin palatal tissue as recently it was recommended to keep 2mm of soft tissue thickness covering the palate to minimize the postoperative pain. Otherwise, necrosis/dehiscence of the flap may happen which was reported to occur frequently for the trap-door approach. Moreover, it is necessary to extend the dissection deeper into the palatal tissues to leave adequate thickness of connective tissue to maintain the vitality of the primary flap which may cause more painful post-operative course.

To overcome these limitations, CTG harvesting with de-epithelialized gingival grafts (DGG) can be executed even in the presence of thin palatal tissues. CTG preparation can be performed more superficially by this approach to obtain collagen-rich connective tissue from Lamina pro- pria of the palatal mucosa. The findings of Zucchelli et al. study support the observation that CTGs which are presumed to have denser connective tissue are comparatively less prone to post-operative shrinkage . According to this assumption, DGG technique may enable to harvest an adequate amount of dense and stable tissue

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years or older. Patients with healthy systemic condition. Buccal recession defects classified as RT-2 recession defects. Clinical indication and/or patient request for recession coverage. O'Leary index less than 20% . No cervical caries or non-carious lesion. No history of periodontal plastic surgery in the affected site

Exclusion Criteria:

Pregnant females. Smokers as smoking is a contraindication for any plastic periodontal surgery Unmotivated, uncooperative patients with poor oral hygiene. Patients with habits that may compromise the longevity and affect the result of the study as alcoholism or para-functional habits.

Overlapping teeth or teeth with abnormal alignment in the dental arch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — the minimum age should be 18 years
Enrollment: 22 (Estimated)
Dates: Start 2019-10-10 (Estimated); Primary Completion 2020-07-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
the distance between the contact point and the top of the papilla | 9 months
  measuring the distance between the contact point and the top of the papilla by graduated William's periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, phd, Study Chair — Cairo University; Hani ElNahass, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
I will check with my study chair

REFERENCES:
- [Result] Aroca S, Keglevich T, Nikolidakis D, Gera I, Nagy K, Azzi R, Etienne D. Treatment of class III multiple gingival recessions: a randomized-clinical trial. J Clin Periodontol. 2010 Jan;37(1):88-97. doi: 10.1111/j.1600-051X.2009.01492.x. Epub 2009 Nov 30. PMID 19968743